CLINICAL TRIAL: NCT06290193
Title: A Prospective Randomized Trial of Acute Normovolemic Hemodilution (ANH) in Patients Undergoing Cytoreductive Surgery for Ovarian Cancer
Brief Title: Study of Acute Normovolemic Hemodilution (ANH) in People With Ovarian Cancer Who Are Having Cytoreductive Surgery
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-392
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Cancer; Fallopian Tube Carcinoma; Ovarian Carcinoma; Peritoneal Carcinoma; Ovarian Cancer Stage IIIC; Fallopian Tube Cancer Stage IIIC; Ovarian Cancer Stage IV; Fallopian Tube Cancer Stage IV; Fallopian Tube Cancer; Peritoneal Cancer
Keywords: ovarian cancer; ovarian carcinoma; ovarian cancer stage IIIC; ovarian cancer stage IV; fallopian tube cancer; fallopian tube carcinoma; fallopian tube cancer stage IIIC; fallopian tube cancer stage IV; peritoneal cancer; peritoneal carcinoma; Acute Normovolemic Hemodilution; Memorial Sloan Kettering Cancer Center; 23-392
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Acute Normovolemic Hemodilution (ANH) Arm (Experimental)
  Interventions: Biological: Acute Normovolemic Hemodilution/ANH
- Standard Intraoperative Management Arm (No Intervention)

INTERVENTIONS:
Biological: Acute Normovolemic Hemodilution/ANH — For participants randomized to ANH, the volume of blood to be removed will be calculated using an established formula, based on preoperative hemoglobin, target hemoglobin after hemodilution, and the patient's estimated blood volume.
  Arms: Acute Normovolemic Hemodilution (ANH) Arm

SUMMARY:
Participants will be scheduled for primary cytoreductive surgery as part of their standard care. Before surgery, participants will be assigned by chance to a study group. Depending on which group they are in, they will receive either acute normovolemic hemodilution/ANH during surgery or standard surgical management during surgery. The researchers think acute normovolemic hemodilution/ANH may decrease the need for allogenic blood transfusion/ABT in people having primary cytoreductive surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years)
* BLOODS score ≥2 as calculated by surgeon
* High preoperative suspicion (or diagnosis) of advanced primary epithelial ovarian, fallopian tube, or primary peritoneal carcinoma (stage IIIC or IV), as determined by CT or MRI of the abdomen/pelvis
* Planned for exploratory laparotomy and primary or interval cytoreductive surgery
* Preoperative hemoglobin concentration ≥10 mg/dl within 45 days of surgery
* Patients scheduled for cytoreductive surgery, with or without other planned procedures o Note: Patients scheduled for only diagnostic laparoscopy should not be included

Exclusion Criteria:

* A history of active coronary artery disease

  o Patients with a history of coronary artery disease will be eligible if they have had a cardiac stress study showing no reversible ischemia and normal LV function within 45 days of surgery.
* A history of cerebrovascular disease
* A history of congestive heart failure
* A history of uncontrolled hypertension
* A history of restrictive or obstructive pulmonary disease
* A history of renal dysfunction (Cr >1.6 mg/dl)
* Abnormal coagulation parameters (INR >1.5 not on coumadin, or platelet count <100,000 mcL)
* Presence of active infection
* Evidence of hepatic metabolic disorder (bilirubin >2 mg/dl, ALT >75 U/L in the absence of biliary tract obstruction)
* Preoperative autologous blood donation within last 30 days or plan to donate autologous blood prior to surgery
* Refusal to accept allogenic or autologous blood transfusion
* Patients scheduled for cytoreductive surgery with planned Hyperthermic Intraperitoneal Chemotherapy (HIPEC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2024-02-23 (Actual); Primary Completion 2029-02-23 (Estimated); Study Completion 2029-02-23 (Estimated)

PRIMARY OUTCOMES:
Comparison of the rate of allogenic red blood cell transfusions between the Acute Normovolemic Hemodilution (ANH) and standard of care arm | up to 30 days from procedure
  The primary objective of this study is to determine if ANH reduces the requirement for allogenic red cell transfusions in patients undergoing primary cytoreductive surgery for ovarian cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Chi, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memoral Sloan Kettering at Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited protocol activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk-Commack (Limited protocol activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited protocol activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All protocol activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org